CLINICAL TRIAL: NCT07127172
Title: GB-PRIME: An Early Feasibility Study of a Precise Robotically Implanted Brain-Computer Interface for the Control of External Devices
Acronym: GB-PRIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuralink Corp (Industry)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other); University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: N1-EFS-006; 354112 (Other: IRAS)
Record Dates: First submitted 2025-07-31; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Tetraplegia/Tetraparesis; Quadriplegia; Quadriplegia/Tetraplegia; Cervical Spinal Cord Injury; Amyotrophic Lateral Sclerosis (ALS); Spinal Cord Injury (Quadraplegia); Spinal Cord Injury; Motor Neuron Disease; Brain Stem Stroke
Keywords: brain computer interface; Neuralink N1 Implant; Neuralink; Robot; tetraparesis; tetraplegia; quadriplegia; ALS; spinal cord injury; Amyotrophic lateral sclerosis; chip; brain chip; External device control; Wireless implant; Neuroprosthetics; SCI; paralysis; motor neuron disease
MeSH Terms: conditions — Quadriplegia; Amyotrophic Lateral Sclerosis; Spinal Cord Injuries; Motor Neuron Disease; Brain Stem Infarctions; Paralysis

STUDY DESIGN:
Intervention Model Description: The study is a pre UKCA/CE, prospective, longitudinal, non-randomized, open-label, single-arm early feasibility study (EFS)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GB-PRIME: Precise Robotically Implanted Brain-Computer Interface (Other): Open label
  Interventions: Device: N1 Implant; Device: R1 Robot

INTERVENTIONS:
Device: N1 Implant — The N1 Implant is a type of implantable brain-computer interface.
Device: R1 Robot — The R1 Robot is a robotic electrode thread inserter that implants the N1 Implant.

SUMMARY:
The GB-PRIME Study is an early feasibility study designed to assess the clinical safety and functionality of the Neuralink N1 Implant and R1 Robot. This study involves participants who have tetraparesis, tetraplegia, or a diagnosis that may lead to these conditions.

The N1 Implant is a wireless, rechargeable device mounted on the skull, connected to electrode threads that are inserted into the brain by the R1 Robot, which is a robotic device specifically designed for this procedure.

ELIGIBILITY:
Inclusion Criteria:

* (a) A diagnosis of a spinal cord injury, brain stem stroke, or other neurological condition causing the participant to be non-ambulant and with bilateral upper limb motor impairment with no expectation of recovery that significantly or completely impairs the participant's ability to manually control a computer, smartphone or tablet with their hands.

OR (b) A diagnosis of Amyotrophic Lateral Sclerosis (ALS) or other progressive neurological condition where the natural history of the disease is well understood and where there is tetraparesis and the expectation in the view of the participants treating neurologist that the disease will progress such that the participant will meet 1a within 1 year of recruitment.

* Life expectancy ≥ 12 months.
* Ability to communicate in English
* Presence of a stable caregiver

Exclusion Criteria:

* Moderate to high risk for serious perioperative adverse events
* Active implanted devices
* Morbid obesity (Body Mass Index > 40)
* History of poorly controlled seizures or epilepsy
* History of poorly controlled diabetes
* Requires magnetic resonance imaging (MRI) for any ongoing medical conditions
* Acquired or hereditary immunosuppression
* Use of smoking tobacco or other tobacco products
* Psychiatric or psychological disorder
* Brain MRI demonstrating hemorrhage, tumor, distorted or adverse anatomy.
* Any condition which, in the opinion of the Investigator, would compromise your ability to safely participate in the study or undergo the implantation procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
The Rate of Device-Related Adverse Events (AE) | 12 months post-implant
The Rate of Procedure-Related Adverse Events (AE) | 12 months post-implant

SECONDARY OUTCOMES:
The Rate of Device-Related Adverse Events (AE) | Up to 48 months post-implant
The Rate of Procedure-Related Adverse Events (AE) | Up to 48 months post-implant
Change in Montreal Cognitive Assessment (MoCA) score during the Primary Study | From baseline to 3-, 6-, 9-, and 12-months post-implantation
  The Montreal Cognitive Assessment (MoCA) is a 30-point scale assessing cognitive function. Scores range from 0 to 30, with higher scores indicating better cognitive performance. Outcome will be reported as change from baseline at each follow-up visit.
Change in Montreal Cognitive Assessment (MoCA) score during the Long-term Follow-up Phase | From baseline to 48-months post-implantation
  The Montreal Cognitive Assessment (MoCA) is a 30-point scale assessing cognitive function. Scores range from 0 to 30, with higher scores indicating better cognitive performance. Outcome will be reported as change from baseline at each follow-up visit.
Change in Patient Health Questionnaire-9 (PHQ-9) score during the Primary Study | From baseline to 1-, 3-, 6-, 9-, and 12-months post-implantation
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item scale used to assess depression severity. Scores range from 0 to 27, with higher scores indicating more severe depressive symptoms. Outcome will be reported as change from baseline at each follow-up visit.
Change in Patient Health Questionnaire-9 (PHQ-9) score during the Long-term Follow-up Phase | From baseline to 48-months post-implantation
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item scale used to assess depression severity. Scores range from 0 to 27, with higher scores indicating more severe depressive symptoms. Outcome will be reported as change from baseline at each follow-up visit.
Change in Generalized Anxiety Disorder-7 (GAD-7) score during the Primary Study | From baseline to 1-, 3-, 6-, 9-, and 12-months post-implantation
  The Generalized Anxiety Disorder 7-item (GAD-7) scale assesses anxiety severity. Scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms. Outcome will be reported as change from baseline at each follow-up visit.
Change in Generalized Anxiety Disorder-7 (GAD-7) score during the Long-term Follow-up Phase | From baseline to 48-months post-implantation
  The Generalized Anxiety Disorder 7-item (GAD-7) scale assesses anxiety severity. Scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms. Outcome will be reported as change from baseline at each follow-up visit.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University College London Hospitals NHS Foundation Trust, London, Greater London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Tyne and Wear

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Neuralink UK Patient Registry — https://neuralink.com/patient-registry/uk/
- See also: Neuralink Website — https://neuralink.com/